CLINICAL TRIAL: NCT02241902
Title: Does Postoperative Pyuria Influence Treatment Outcomes After Photoselective Vaporization of the Prostate (PVP)?: A Short-term Serial Follow-up Study
Brief Title: Impact of Postoperative Pyuria on Treatment Outcomes After PVP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: DongGuk University (Other)
Responsible Party: Principal Investigator, Min Chul Cho, Assistant professor, DongGuk University
Other Study IDs: MCho1
Record Dates: First submitted 2014-09-13; First posted 2014-09-16 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Prostatic Hyperplasia; Pyuria
MeSH Terms: conditions — Prostatic Hyperplasia; Pyuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- No pyuria
- Persistent pyuria

SUMMARY:
The aim of this study was to identify serial changes in the incidence of postoperative pyuria after the Photoselective Vaporization of the Prostate (PVP), to determine whether the presence of postoperative pyuria could be correlated with surgical outcomes after surgery and to identify predicting factors that influence on persistent pyuria after the PVP.

ELIGIBILITY:
Inclusion Criteria:

* men who underwent photoselective vaporization (PVP) using 80 watt potassium-titanyl-phosphate (KTP) laser or 120 watt high-power-system (HPS) laser for benign prostatic hyperplasia refractory to medical treatment
* sterile urine on urinalysis and urine culture before surgery
* absence of indwelling urethral catheter before surgery

Exclusion Criteria:

* previous diagnosis of prostate carcinoma or bladder cancer
* co-existence of urinary stone
* any antibiotic treatment within 2-weeks before surgery

Ages: 40 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: men who underwent photoselective vaporization (PVP) using 80 watt potassium-titanyl-phosphate (KTP) laser or 120 watt high-power-system (HPS) laser for benign prostatic hyperplasia refractory to medical treatment
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Change in the subtotal storage symptoms score of the International Prostate Symptom Score (IPSS) | 1-week, and 1-, 3- and 6-months after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Min Chul Cho, M.D., Ph.D., Principal Investigator — DongGuk University
Locations (1):
- Dongguk University ilsan Hospital, Goyang-si, Gyeonggi-do, South Korea